CLINICAL TRIAL: NCT06410989
Title: Relating Ankle Impairments to Walking Ability for Characterization of Sensorimotor Function in Individuals With Chronic Stroke
Brief Title: Evaluation of Sensorimotor Ankle Impairments in Chronic Stroke
Status: Not yet recruiting | Type: Observational
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Jose Pons, Principal Investigator, Shirley Ryan AbilityLab
Other Study IDs: STU00219274
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: Robotic Rehabilitation; Sensorimotor function; Proprioception; Motor Control; Ankle Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Chronic patients post-stroke: Patients post-stroke, age 40-80, with a unilateral supratentorial ischemic or hemorrhagic stroke
- Healthy Individuals: Healthy adults, age 40-80, without neurological disorders

SUMMARY:
The purpose of this study is to capture sensorimotor ankle function in a chronic stroke population through validation of novel, experimental metrics and their comparison with established, clinical measures of function. For this purpose, the researchers will evaluate various single-joint, impairment-level measures such as visuomotor tracking performance and proprioception as well as functional-level measures including spatiotemporal gait (e.g., gait speed and stride length/time) and standardized clinical scales. This study will be carried out in chronic stroke patients as well as age-matched healthy controls. Results will help the researchers identify more quantitative metrics that can be used to monitor and rehabilitate sensorimotor function following stroke.

DETAILED DESCRIPTION:
The purpose of this study is to capture sensorimotor ankle function in a chronic stroke population through validation of novel, experimental metrics and their comparison with established, clinical measures of function. Target populations will perform various single-joint ankle tasks (i.e., dorsiflexion and plantarflexion), assessing the quality of their movements during visuomotor tracking, goal-directed movements and unilateral/bilateral tests of joint position and force sense. Collecting these data will delineate which measures of ankle function are specific to chronic stroke, as well as sensitivity to the severity of stroke, assessed via the Fugl-Meyer Assessment for the Lower Extremity. In addition, the investigators will determine the relationship between deficits in proprioception and assessments which integrate multiple feedback modalities (i.e., proprioception, motor control and vision) to assess the role of peripheral sensory feedback in performing ankle movements post-stroke. The investigators will correlate measures of ankle impairment to clinical scales commonly used in physical therapy. As a first step, the investigators will directly compare these ankle measures to clinical tests of ankle sensation and motor control to demonstrate improvements in assessment sensitivity with this method. Furthermore, the investigators will correlate these ankle measures with clinical measures of lower-limb function during ambulatory and balance tasks, to better understand the contribution of ankle impairments to dynamic, multi-joint activities in chronic stroke.

ELIGIBILITY:
Inclusion criteria

* 40 - 80 years of age, inclusive
* Normal hearing and vision, can be corrected
* No skin allergies to adhesive material, conductive paste, or silver
* Ability to walk >10m independently on level ground without an assistive device or bracing
* Able to understand and give informed consent
* Able to understand and speak English

Inclusion criteria specific for healthy participants:

* No neurological disorders
* Absence of pathology that could cause abnormal movements of extremities (e.g., epilepsy, stroke, marked arthritis, chronic pain, musculoskeletal injuries)

Inclusion criteria specific for participants post-stroke:

* Unilateral, supratentorial ischemic or hemorrhagic stroke ≥ six months prior
* Minimum activation against gravity for dorsiflexion and plantarflexion, equivalent to a Manual Muscle Test (MMT) score of ≥ +2
* Self-selected walking speed is less than 1.2 m/s

Exclusion criteria

* Cognitive limitations that would prevent playing games
* Adults unable to consent, pregnant women, children, or prisoners
* Infection, wounds, or graft sites on lower limbs
* History of sustained non-prescribed drug use or substance abuse (as reported by subject; current nicotine use is allowed)
* History of peripheral nerve injury
* Severe hip, knee, or ankle arthritis
* Recent fracture or osteoporosis (as reported by subject)
* Bone or joint instability in the lower limb
* Severe pain syndromes affecting any part of the lower limbs
* Fixed contractures affecting the lower limbs
* Medical (cardiac, renal, hepatic, oncological) or psychiatric disease that would interfere with study procedures
* Inability or unwillingness to perform study-required activities
* Prior neurosurgical procedures

Exclusion criteria specific for healthy participants:

- Any neurological diseases (e.g., stroke, Parkinson's disease or other neurodegenerative disorder, severe dementia, brain injury, spinal cord injury, multiple sclerosis, or cancer of the central nervous system)

Exclusion criteria specific for participants post-stroke:

* Co-existence of other neurological diseases (e.g., Parkinson's disease or other neurodegenerative disorder, severe dementia, brain injury, spinal cord injury, multiple sclerosis, or cancer of the central nervous system)
* Botox (botulinum toxin) injection to lower limbs within the prior 3 months
* Significant spasticity or contracture in the lower limbs (Modified Ashworth Scale score of 4)
* Severe aphasia
* Significant loss of sensation in the lower limbs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chronic patients post-stroke and healthy individuals as controls
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Sensation and voluntary control of the ankle, quantified by spatiotemporal errors during visuomotor tracking and matching tasks using a robotic ankle device | Assessment during a single 2-hour study visit
  Ankle function will be measured with a robotic device while the participant performs various dorsiflexion and plantarflexion movements to evaluate their ankle motor control and proprioception. For the visuomotor tracking tasks, participants will repetitively perform a specified movement, guided by visual feedback of their own input and a target movement to follow. In the matching tasks, participants will be asked to reproduce different ankle configurations (i.e., maintaining a target force or position) based on their memory of previous configurations. In both tasks, errors between the target movement and the participant's movement will be compared between chronic stroke and age-matched cohorts to characterize ankle deficits associated with stroke.

SECONDARY OUTCOMES:
Correlation between spatiotemporal ankle control and clinical measurement of ankle control | Assessment during a single 2-hour study visit
  The Manual Muscle Test (MMT) will be used as a measure of voluntary ankle control and compared to the spatiotemporal errors defined in the primary outcome measures section.
Correlation between spatiotemporal ankle control and spatiotemporal gait measures during overground walking | Assessment during a single 2-hour study visit
  The 10 meter walk test will be used to measure the participant's comfortable walking speed and spatiotemporal gait parameters (i.e., stride length and stride time); these measures will be compared to the spatiotemporal errors defined in the primary outcome measures section.
Correlation between spatiotemporal ankle control and gait endurance | Assessment during a single 2-hour study visit
  The 6 minute walk test will be used to measure the participant's endurance during gait and will be compared to the spatiotemporal errors defined in the primary outcome measures section.
Correlation between spatiotemporal ankle control and clinical scales of sensation | Assessment during a single 2-hour study visit
  The Monofilament test will be used to measure the participant's touch sensitivity at the ankle and will be compared to the spatiotemporal errors defined in the primary outcome measures section.

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Pons, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No